CLINICAL TRIAL: NCT00687908
Title: Efficacy and Safety Comparison of Adapalene 0.1% / Benzoyl Peroxide 2.5% Gel Versus Adapalene 0.1% / Benzoyl Peroxide 2.5% Gel Vehicle Gel as a 6-month Acne Maintenance Treatment
Brief Title: Adapalene-Benzoy Peroxide (BPO) Gel in the Treatment of Acne Vulgaris as a 6-month Maintenance
Acronym: ACCESS II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Jean-Charles DHUIN Clinical Trial Manager, Galderma
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RD.03.SPR.29075
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Results first posted 2010-09-24 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2010-09

CONDITIONS: Acne
Keywords: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene; Benzoyl Peroxide; Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Adapalene 0.1% / Benzoyl Peroxide 2.5% Gel once daily
  Interventions: Drug: Adapalene 0.1% / Benzoyl Peroxide 2.5% Gel
- 2 (Placebo Comparator): Vehicle Gel once daily
  Interventions: Drug: Vehicle Gel

INTERVENTIONS:
Drug: Adapalene 0.1% / Benzoyl Peroxide 2.5% Gel — Topical Gel to the face, once daily in the evening for 24 weeks.
  Other Names: Adapalene-BPO gel
  Arms: 1
Drug: Vehicle Gel — Topical Gel to the face, once daily in the evening for 24 weeks.
  Arms: 2

SUMMARY:
The purpose of this study is to demonstrate the efficacy of Adapalene 0.1% /Benzoyl Peroxide 2.5% Gel compared to its Vehicle Gel as an acne maintenance treatment in Subjects previously treated with Adapalene-BPO Gel or Adapalene-BPO Vehicle Gel both associated with Doxycycline Hyclate 100 mg. The safety of the two investigational treatments will also be assessed.

DETAILED DESCRIPTION:
This study is a follow-up to RD.03.SPR.29074 - ACCESS I / NCT00688064 - "Adapalene-BPO Gel Associated With Doxycycline 100 mg in the Treatment of Severe Acne Vulgaris"

ELIGIBILITY:
Inclusion Criteria:

* Subjects who completed the previous study (RD.03.SPR29074 - NCT00688064)and had obtained at least a good Improvement (Grade, 0, 1, 2 or 3)

Exclusion Criteria:

* Female Subjects who are pregnant, nursing or planning a pregnancy during the study
* Subjects who foresee intensive UV exposure during the study (mountain sports, UV radiation, sunbathing, etc).

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 243 (Actual)
Dates: Start 2008-11; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane Thiboutot, MD, Principal Investigator — Penn State College of Medicine, Hershey, PA
Locations (33):
- United States (27):
  - Galderma Investigational Site, San Diego, California
  - Galderma Investigational Site, Denver, Colorado
  - Galderma Investigational Site, Longmont, Colorado
  - Galderma Investigational Site, Miami, Florida
  - Galderma Investigational Site, Snellville, Georgia
  - Galderma Investigational Site, Chicago, Illinois
  - Galderma Investigational Site, Evansville, Indiana
  - Galderma Investigational Site, Overland Park, Kansas
  - Galderma Investigational Site, Louisville, Kentucky
  - Galderma Investigational Site, Detroit, Michigan
  - Galderma Investigational Site, Fort Gratiot, Michigan
  - Galderma Investigational Site, Fridley, Minnesota
  - Galderma Investigational Site, Omaha, Nebraska
  - Galderma Investigational Site, Albuquerque, New Mexico
  - Galderma Investigational Site, Stony Brook, New York
  - Galderma Investigational Site, Winston-Salem, North Carolina
  - Galderma Investigational Site, Warren, Ohio
  - Galderma Investigational Site, Hazleton, Pennsylvania
  - Galderma Investigational Site, Hershey, Pennsylvania
  - Galderma Investigational Site, Simpsonville, South Carolina
  - Galderma Investigational Site, Arlington, Texas
  - Galderma Investigational Site, Austin, Texas
  - Galderma Investigational Site, College Station, Texas
  - Galderma Investigational Site, Houston, Texas
  - Galderma Investigational Site, Lubbock, Texas
  - Galderma Investigational Site, San Antonio, Texas
  - Galderma Investigational Site, Webster, Texas
- Canada (4):
  - Galderma Investigational Site, Barrie, Ontario
  - Galderma Investigational Site, North Bay, Ontario
  - Galderma Investigational Site, Windsor, Ontario
  - Galderma Investigational Site, Québec, Quebec
- Puerto Rico (2):
  - Galderma Investigational Site, Aibonito
  - Galderma Investigational Site, Carolina

REFERENCES:
- See also: Related Info — http://galderma.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 12 NOV 2008 to 09 FEB 2009 in thirty-four centers (29 in the USA and 5 in Canada) public or private practices. Twenty-four USA centers and four Candadian centers used a central IRB, and the others used a local IRB.
Groups:
- Adapalene-BPO: Adapalene 0.1% / Benzoyl Peroxide 2.5% Gel
- Vehicle: Vehicle Gel
Period: Overall Study
Arm/Group | Adapalene-BPO | Vehicle
Started | 123 | 120
Completed | 105 | 78
Not Completed | 18 | 42

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adapalene-BPO | Vehicle | Total
Number analyzed (Participants) | 123 | 120 | 243
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 76 | 84 | 160
  Between 18 and 65 years | 47 | 36 | 83
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.1 (5.89) | 18.2 (5.23) | 18.6 (5.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 53 | 111
  Male | 65 | 67 | 132
Region of Enrollment [Number; unit: participants]
  United States | 84 | 79 | 163
  Puerto Rico | 13 | 13 | 26
  Canada | 26 | 28 | 54

OUTCOME MEASURES:

1. Primary Outcome: Maintenance Success for Total Lesions at Week 24
Description: Maintenance success for total lesions at Week 24 is defined as the percentage of subjects maintaining at least 50 percent of the improvement obtained with prior combination therapy, in terms of total lesion counts.
Time Frame: Week 24
Population: ITT - Worst-case (Any missing data at Week 24 is considered as a failure)
Measure: Number; unit: percent of subjects
Arm/Group | Adapalene-BPO | Vehicle
Number analyzed (Participants) | 123 | 120
percent of subjects | 78.9 | 45.8

2. Secondary Outcome: Maintenance Success for Inflamatory Lesions at Week 24
Description: Maintenance success for inflamatory lesions at Week 24 is defined as the percentage of subjects maintaining at least 50 percent of the improvement obtained with prior combination therapy, in terms of inflamatory lesion counts.
Time Frame: Week 24
Population: ITT - Worst-case (Any missing data at each visit is considered as a failure, except where maintenance rate of both previous and following visits are success)
Measure: Number; unit: percent of subjects
Arm/Group | Adapalene-BPO | Vehicle
Number analyzed (Participants) | 123 | 120
percent of subjects | 78 | 48.3

3. Secondary Outcome: Maintenance Success for Non-inflammatory Lesions at Week 24
Description: Maintenance success for non-inflamatory lesions at Week 24 is defined as the percentage of subjects maintaining at least 50 percent of the improvement obtained with prior combination therapy, in terms of non-inflamatory lesion counts.
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: percent of subjects
Arm/Group | Adapalene-BPO | Vehicle
Number analyzed (Participants) | 123 | 120
percent of subjects | 78 | 43.3

4. Secondary Outcome: Investigator Global Assessment (IGA) Maintenance Success at Week 24
Description: IGA maintenance success is defined as the percentage of subjects with IGA grade inferior or equal to Baseline IGA grade.
  IGA grade:
  0 Clear:Residual hyperpigmentation & erythema may be present
  1. Almost Clear:A few scattered comedones & a few small papules.
  2. Mild:Some comedones & some papules and pustules. No nodules present
  3. Moderate:Many comedones, papules & pustules. One nodule may be present
  4. Severe:Covered with comedones, numerous papules & pustules & few nodules & cysts may be present
  5. Very severe:Highly inflammatory acne covering the face; with nodules & cysts present
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Number; unit: percent of subjects
Arm/Group | Adapalene-BPO | Vehicle
Number analyzed (Participants) | 123 | 120
percent of subjects | 70.7 | 34.2

5. Secondary Outcome: Percent of Subjects With Adverse Events
Description: All participants with events were measured for that particular Outcome Measure and not only the events with a frequency threshold above 2 percent
Time Frame: Up to 24 weeks
Measure: Number; unit: percent of subjects
Arm/Group | Adapalene-BPO | Vehicle
Number analyzed (Participants) | 123 | 120
percent of subjects | 41.5 | 29.2

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Adapalene-BPO | Vehicle
Serious Adverse Events (participants affected / at risk) | 1/123 | 1/120
Other Adverse Events (participants affected / at risk) | 43/123 | 27/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adapalene-BPO (N=123) | Vehicle (N=120)
Bipolar disorder (Nervous system disorders) | 1 (1) | 0 (0)
Pilonidal abscess (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adapalene-BPO (N=123) | Vehicle (N=120)
Headache (Nervous system disorders) | 5 (5) | 3 (3)
Influenza (Infections and infestations) | 4 (4) | 1 (1)
Nasopharyngitis (Infections and infestations) | 8 (10) | 12 (12)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Pharyngitis (Infections and infestations) | 4 (4) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 4 (4) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (3)
Pyrexia (General disorders) | 4 (4) | 1 (1)
Sinusitis (Infections and infestations) | 4 (4) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any intent of the investigator to publish or disclose in any way the information requires the sponsor's prior written approval. The investigator shall provide their draft of such publication to sponsor for review and approval at least 2 months prior to the date of the intended publication. Sponsor shall have the absolute right to determine whether information may be published by the investigator.